CLINICAL TRIAL: NCT06004869
Title: Incorporating Ecological Momentary Assessment and Intervention Into Cognitive Behavioural Therapy for Insomnia Using mHealth and Wearable Technologies: A Pilot Randomised Controlled Trial
Brief Title: Incorporating EMA and EMI Into CBT-I Using mHealth and Wearable Technologies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSY031
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Insomnia
Keywords: ecological momentary intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ecological Momentary Assessment; Methods; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMA/I CBT-I group (Experimental): The participants allocated to the EMI/A CBT-I group will receive 6 weeks of smartphone-based CBT-I for approximately 1 hour per week. The EMA feature will capture the participant's momentary ratings of experiences to support therapeutic decision making. The trained therapist will prescribe EMI, provide personalised sleep advice, and adjust the treatment by dynamically adapting real-time rest-activity assessments collected using EMA and wearable devices. The participants will receive tailored moment-specific feedback from therapists when daytime symptoms are indicated. Therapists will also monitor the relationship between daytime symptoms (EMA app) and the sleep-wake pattern (wearables).
  Interventions: Behavioral: Ecological momentary assessments/interventions with cognitive behavioural therapy for insomnia (EMA/I CBT-I)
- Pure self-help CBT-I group (Active Comparator): The participants in the pure self-help CBT-I group will receive 6 weeks of self-help CBT-I without EMA/I and therapist support. The CBT-I content will be identical to the content used in the EMI/A CBT-I group.
  Interventions: Behavioral: Self-help cognitive behavioural therapy for insomnia
- Care as usual (No Intervention)

INTERVENTIONS:
Behavioral: Ecological momentary assessments/interventions with cognitive behavioural therapy for insomnia (EMA/I CBT-I) — an integrated system based on an existing multicomponent cognitive behavioural therapy for insomnia (CBT-I) and EMA app
  Arms: EMA/I CBT-I group
Behavioral: Self-help cognitive behavioural therapy for insomnia — An mobile app that delivers CBT-I content.
  Arms: Pure self-help CBT-I group

SUMMARY:
This study will be a randomised controlled trial to investigate an integrated platform that incorporates ecological momentary assessments/interventions (EMA/I) into cognitive behavioural therapy for insomnia (CBT-I) using mHealth and wearable technology. The intervention is a promising prospect to address current challenges in the context of sleep medicine to provide real-time and real-world intervention with accuracy, low cost, and easy accessibility.

DETAILED DESCRIPTION:
It will be a randomised, assessor-blind controlled trial embedding both outcome and process evaluation, of the EMA/I CBT-I in conjunction with wearable sensors. The outcome evaluation will examine the treatment effect of EMA/I CBT-I compared with care-as-usual (CAU), whilst process evaluation will enhance the understanding of the causal assumptions that underpin EMA/I CBT-I to inform policy and clinical practice. 60 eligible participants will be randomly assigned to the EMA/I CBT-I group and CAU in a 1:1 allocation ratio. The participants in the EMA/I CBT-I group will receive 6 weeks of smartphone-based EMA/I CBT-I supported by a therapist. The trained therapist will prescribe EMI, provide personalised sleep advice, and adjust the treatment by dynamically adapting real-time rest-activity assessments collected using EMA and wearable devices. Assessments will be managed by an independent assessor (a research assistant) who is blind to group allocation at baseline, week 7 (1 week after treatment), and week 18 (12 weeks after treatment). The proposed study will follow the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) and will be registered on ClinicalTrials.gov to ensure compliance with study design and results reporting requirements. The treatment will be provided free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents at least 18 years of age;
2. able to read Chinese and type in Chinese or English;
3. meet the DSM-5 diagnostic criteria of insomnia disorder (difficulty initiating and/or maintaining sleep or early morning awakening, alongside clinically significant daytime impairment) based on the Brief Insomnia Questionnaire (BIQ), a diagnostic tool validated by the team;
4. have an Insomnia Severity Index (ISI) score of at least 10 indicating clinical-level insomnia;
5. have adequate opportunity and circumstances for sleep to occur;
6. have an Internet-enabled mobile device (iOS or Android operating system), and
7. are willing to provide informed consent.

Exclusion Criteria:

To mimic real-world settings, a less stringent set of exclusion criteria will be adopted.

1. A Beck Depression Inventory (BDI-II) Item 9 score of at least 2 indicating a current moderate suicidal risk that requires active crisis management (referral information to professional services will be provided to those with serious suicidal risk);
2. involvement in CBT-I in the past 6 months;
3. a history of severe mental illness (e.g., bipolar disorder, psychotic disorder);
4. major medical or neurocognitive disorders or side effects of medication that contribute significantly to insomnia or make participation infeasible based on the team's clinical experience;
5. other untreated sleep disorders, including narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS)/periodic leg movement disorder (PLMD) based on the cut-off scores (≥7 on narcolepsy; ≥15 on OSA; ≥7 on RLS/PLMD) in SLEEP-50;
6. taking over-the-counter medication or psychotropic drugs that target insomnia within 2 weeks prior to the baseline assessment; and
7. shift work, pregnancy, family or other commitments that interfere with regular sleep-wake patterns.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Insomnia Severity Index (ISI) | Baseline, Immediate post-treatment, 12-week follow up
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5- point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeable impairment attributed to the sleep problem, and level of distress caused by the sleep problem.

SECONDARY OUTCOMES:
Changes in the Pittsburgh Sleep Quality Index (PSQI-19) | Baseline, Immediate post-treatment, 12-week follow up
  The PSQI-19 is a 19-item questionnaire used for measuring and identifying the quality of sleep. It provides a measure of global sleep quality, including sleep latency, sleep duration, habitual sleep efficiency and sleep disturbances.
Changes in 7-Day Consensus Sleep Diary | Baseline, Immediate post-treatment, 12-week follow up
  The standardized sleep diary records sleep-onset latency (SOL; min), wake after sleep onset (WASO; min), total wake time (TWT; min), total sleep time (TST; min), time in bed (TIB; min), etc.
Changes in Hospital Anxiety and Depression Scale (HADS) | Baseline, Immediate post-treatment, 12-week follow up
  A 14-item self-rating scale that measures anxiety and depression in both hospital and community settings. It is divided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items. It is for screening purposes and is not meant to be a diagnostic tool. HADS scores of 8-10, 11-14, and 15-21 represent mild, moderate, and severe anxiety and depression separately.
Changes in Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) | Baseline, Immediate post-treatment, 12-week follow up
  The DBAS is a 16-item questionnaire used to assess sleep-related cognitions.
Changes in the Epworth Sleepiness Scale (ESS) | Baseline, Immediate post-treatment, 12-week follow up
  The ESS is an 8-item scale designed to evaluate overall daytime sleepiness.
Changes in Multidimensional Fatigue Inventory (MFI) | Baseline, Immediate post-treatment, 12-week follow up
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Scores on each subscale range from 4 to 20, with higher scores indicating greater fatigue.
Changes in Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, Immediate post-treatment, 12-week follow up
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state).
Changes in Sheehan Disability Scale (SDS) | Baseline, Immediate post-treatment, 12-week follow up
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Changes in Credibility-Expectancy Questionnaire (CEQ) | Baseline, Immediate post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Changes in Insomnia Treatment Acceptability Scale (ITAS) | Baseline, Immediate post-treatment
  The 8-item Insomnia Treatment Acceptability Scale (ITAS) may examine treatment acceptability. Respondents would score each item from 0 (not at all acceptable) to 4 (very acceptable) to rate if the rationale made sense, how acceptable the treatment was for them, suitability for their sleep problem, and expected effectiveness for their sleep problem.